CLINICAL TRIAL: NCT05415280
Title: Impact of Mindfulness Based Intervention on the COVID-19 Related Distress and Mobile Addiction During Pandemic: A Randomized Control Trails
Brief Title: Mindfulness Based Intervention on the COVID-19 Related Distress and Mobile Addiction
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fatima Jinnah Women University (Other)
Responsible Party: Principal Investigator, Zia-un-nisa, Principal Investigator, Fatima Jinnah Women University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MBSR
Record Dates: First submitted 2022-02-24; First posted 2022-06-13 (Actual); Last update posted 2022-06-14 (Actual); Status verified 2022-06

CONDITIONS: Psychological Stress
Keywords: psychological stress mobile phone addiction
MeSH Terms: conditions — Stress, Psychological | interventions — Mindfulness-Based Stress Reduction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness based stress reduction (Experimental): mindfulness based stress reduction intervention was used to treat psychological and addiction problems of the individuals
  Interventions: Behavioral: Mindfulness Based stress reduction
- Relaxation Exercise (Other): the control group was provided with the relaxation technique.
  Interventions: Behavioral: Mindfulness Based stress reduction

INTERVENTIONS:
Behavioral: Mindfulness Based stress reduction — The aim of the psychological intervention to reduce the mental health problems of the participants.

SUMMARY:
The interventional study would be conducted to investigate the efficacy of mindfulness based intervention in order to treat psychological stress(anxiety, depression, and stress related COVID-19), and mobile phone addiction during COVID-19 pandemic.

DETAILED DESCRIPTION:
In the current study the data was collected from the young adults (age range 19-35 years). The high scorer from the sample selected from the participants in both control and experimental groups. furthermore, the mindfulness based stress reduction intervention was given to the experimental group. The mindfulness based stress reduction intervention comprised eight weeks period. After the provision of intervention the data for the second phase would be collected.

ELIGIBILITY:
Inclusion Criteria:

* The participants fulfil the age criteria, students from public and private universities, and provided signed informed consent.

Exclusion Criteria:

* Participant suffering from chronic physical or psychological disorder. In addition participant who experience death of loved ones during COVID-19 pandemic.

Ages: 19 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-08-01 (Estimated); Primary Completion 2022-10-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
COVID-19 related Stress | 35 minutes
  COVID-19 related stress scale(<5 minimum, >72 Maximum)
anxiety and depression | 15 minutes
  hospitalized anxiety and depression scale (<7 minimum, >21 Maximum)

SECONDARY OUTCOMES:
mobile phone addiction | 35 minutes
  smartphone addiction scale (33 minimum, 198maximum)

CONTACTS AND LOCATIONS:
Overall Officials: zia-un Nisa, Principal Investigator — assisstant professor
Locations (1):
- Zia-Un Nisa, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No
The investigator has not plan to share data without taking permission from the study participants.